CLINICAL TRIAL: NCT04247113
Title: Assessing the Feasibility and Acceptability of a Parent-Based Intervention to Reduce the Risk of Obesity in Children of Weight Loss Surgery Patients
Brief Title: Parent-Based Intervention Following a Weight Loss Surgery
Acronym: PBP-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, James Dale Lock, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 36281
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Obesity, Childhood
Keywords: bariatric surgery; Parent-based prevention
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBP-B (Experimental): Parent-based Prevention following a Bariatric Surgery (PBP-B) is a 6-session parent-based program designed to guide parents who have undergone a weight loss surgery and their partners in developing healthy eating habits in their children
  Interventions: Behavioral: Parent-based prevention following bariatric surgery

INTERVENTIONS:
Behavioral: Parent-based prevention following bariatric surgery — PBP-B is an adapted version of Parent-Based Prevention (PBP), an innovative approach with demonstrated efficacy in targeting the familial effects of parents with eating disorders on their young children's healthy behaviors. PBP-B addresses the parental cognitions and behaviors that putatively increase the risk for maladaptive outcomes in their children.

SUMMARY:
Prevention and early intervention are the most effective methods for influencing eating habits. This study helps fulfill the Department of Psychiatry's missions of clinical innovation and advancing science. Findings will inform future clinical practice, improve the care provided to patients in their important role as parents, and foster interdisciplinary collaborations.

DETAILED DESCRIPTION:
Morbid obesity is both highly heritable and affected by environmental factors. The child of a parent undergoing a weight-loss surgery (PWLS) is at especially high risk of obesity. The most effective approach to reducing the risk of childhood obesity is a parent-based program. However, adherence remains a challenge, largely due to lack of tailored interventions. Typical interventions are not individualized to target the unique characteristics of the family nor timed to be delivered when the family is geared for change. Parent-Based Prevention following a bariatric surgery (PBP-B) is a novel targeted intervention that focuses on parental behaviors important for developing healthy eating and lifestyle behaviors in young children. PBP-B personalizes treatment goals through a focused parent-based approach that includes a family meal. Additionally, PBP-B is timed to capitalize on the Halo Effect period, in which the BMIs of the family members of the person undergoing weight loss surgery reduce spontaneously, yet only temporarily.

This study will investigate whether PBP-B is feasible, acceptable, and associated with improvement in short-term outcomes that predict long term risks of obesity (e.g., parental feeding practices, child eating behaviors, child physical activity levels, and child sleep hours). Ten adults who had weight loss surgery and are the parents of one or more children aged 1-10 will receive PBP-B (with their partners, unless they are single parents). This study will collect important pilot data that will inform the design of future adequately powered studies to test ways to reduce the likelihood of adult obesity in children of a parent who had weight loss surgery.

ELIGIBILITY:
Inclusion Criteria:

* The biological parent of a child between 1-10 years of age.
* Has undergone a weight loss surgery.

Exclusion Criteria:

* Current medical condition necessitating more intensive care to manage symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting parents who have undergone a bariatric surgery | Up to 18 months
  Number of eligible participants that agree to participate in the study
Acceptability of the intervention | Week 8
  Client Satisfaction Questionnaire score at end of treatment

SECONDARY OUTCOMES:
Parental feeding practices | Baseline and Week 8
  Change scores of the Child Feeding Questionnaire from baseline to end of treatment
Child eating behaviors | Baseline and Week 8
  Change scores of the Children's Eating Behavior Questionnaire from baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Safer, MD, Principal Investigator — Stanford University; Shiri Sadeh-Sharvit, PhD, Principal Investigator — Stanford University; James Lock, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No